CLINICAL TRIAL: NCT03368612
Title: Comparative Study Between the AirGoTM System and Standard Tests in the Assessment of the Respiratory Function
Acronym: AirGoTM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale Santa Croce-Carle Cuneo (Other)
Responsible Party: Principal Investigator, Andrea Antonelli, Principal Investigator, MD, Ospedale Santa Croce-Carle Cuneo
Other Study IDs: A.O. S. Croce e Carle di Cuneo
Record Dates: First submitted 2017-11-14; First posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Respiration Disorders
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Electronic evaluation system — spirometry, plethysmography, cardiopulmonary exercise test
Other: Electronic evaluation system — AirGo recording
  Other Names: AirGoTM System

SUMMARY:
The study aims at evaluating the AirGoTM system's performance, as compared to standard pulmonary function tests.

DETAILED DESCRIPTION:
Primary endpoint:

• To test the AirGoTM system's respiratory rate recording accuracy at rest and during physical exercise, as compared to standard tests.

Secondary endpoints:

* To test the accuracy of the AirGoTM system's derived respiratory parameters (tidal volume, minute ventilation, Tiffeneau-Pinelli index, FEV1 and VO2max) at rest and during physical exercise, as compared to standard tests.
* To test comfort and subjects' compliance with the AirGoTM system during long term recording (24 hours).

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker healthy volunteers,
* Able to perform a routine respiratory function test (spirometry and cardiopulmonary exercise testing),
* aged between 18 and 75 years,
* who signed a written informed consent.

Exclusion Criteria:

* Present cardiac comorbidities (eg. coronary artery disease, heart failure, arrhythmias);
* History of coronary artery disease or heart failure;
* Respiratory comorbidities (eg. asthma, chronic obstructive disease, sleep apnoea, lung interstitial disease);
* Pregnancy;
* Former smoker of >5 p/y;
* Severe trauma or major surgery in the last year;
* Chest pain;
* Obesity (BMI >30).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-09-22 (Actual); Primary Completion 2019-09-22 (Estimated); Study Completion 2019-09-22 (Estimated)

PRIMARY OUTCOMES:
respiratory rate | 4 minutes
  number of respiratory cycles completed in one minute

SECONDARY OUTCOMES:
tidal volume | 4 minutes
  volume of air moved during a single respiratory cycle (inspiration and expiration) during normal breathing (in ml)

CONTACTS AND LOCATIONS:
Locations (1):
- A.O. S. Croce E Carle Di Cuneo, Cuneo, Italy

IPD SHARING:
Plan to Share IPD: No